CLINICAL TRIAL: NCT04467281
Title: A Diagnostic Study of CD38-Targeted ImmunoPET of Myeloma: Phase 2 Trial of Clinical Applications
Brief Title: A Study of PET/CT Scans With the Radioactive Tracer 89Zr-DFO-Daratumumab in People With Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution and study is being transferred.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-098
Record Dates: First submitted 2020-07-02; First posted 2020-07-13 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: CD38-Targeted ImmunoPET; 20-098
MeSH Terms: conditions — Multiple Myeloma | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: This will be a phase II clinical trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-DFO-daratumumab PET/CT (Experimental): Pre treatment evaluation: 1) Standard of Care (SoC) labs, imaging, blind bone marrow biopsy. 2) Baseline research 89 Zr DFO daratumumab PET/CT 3) Possible biopsy of 89 Zr DFO daratumumab avid lesion Treatment: Daratumumab containing combination therapy (up to 12 cycles, 4 weeks/cycle). SoC labs, imaging, and blind bone marrow biopsies until complete response (CR) is suspected or 12 cycles are completed.
  Post treatment evaluation:1) SoC labs, imaging, and blind bone marrow biopsy 2) SoC minimal residual disease (MRD) analysis by next generation sequencing 3) Follow up research 89 Zr DFO daratumumab PET/CT 4) Possible biopsy of 89 Zr DFO daratumumab avid lesion
  Interventions: Drug: 89Zr-DFO-daratumumab; Diagnostic Test: PET/CT

INTERVENTIONS:
Drug: 89Zr-DFO-daratumumab — Patients will undergo 89Zr-DFO-daratumumab PET/CT once before standard of care therapy and once again afterward, for a total of two research scans.
Diagnostic Test: PET/CT — Patients will undergo 89Zr-DFO-daratumumab PET/CT once before standard of care therapy and once again afterward, for a total of two research scans.

SUMMARY:
The purpose of this study is to see if using the radioactive tracer 89Zr-DFO-daratumumab with PET/CT scans is a practical and effective way to view and monitor multiple myeloma in participants before and during their treatment with daratumumab. We also want to see if 89Zr-DFO-daratumumab PET/CT scans can predict a participant's response to therapy, and if they can better locate any leftover disease following treatment compared to the standard imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Histologically/immunohistochemistry-confirmed CD38-positive multiple myeloma
* At least one tumor lesion on CT, MRI, or FDG PET/CT within 90 days of protocol enrollment
* ECOG performance status 0 to 2
* Participant is capable of having an informed consent discussion (Legally Authorized Representatives are not permitted to sign on a participant's behalf).

Exclusion Criteria:

* Life expectancy < 12 months
* Pregnancy or lactation
* Patients who cannot undergo PET/CT scanning because of weight limits. PET/CT scanners may not be able to function with patients over 450 pounds.
* History of anaphylactic reaction to humanized or human antibodies.
* Previous treatment with daratumumab. Previous treatment with other myeloma therapies will be allowed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
number of patient's with positive tumors | 1 year
  Uptake of FDG PET/CT

SECONDARY OUTCOMES:
assess if tumor uptake of 89Zr-DFO-daratumumab predicts response to daratumumab/lenalidomide therapy | 1 year
  The response will be defined using IMWG criteria as complete or partial response; stable disease and progressive disease will be considered as non-response.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Mayerhoefer, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm